CLINICAL TRIAL: NCT02279498
Title: A Phase 3, Randomized, Open-Label, Assessor-Blind, Noninferiority, Active-Comparator Study Evaluating the Efficacy and Safety of Liprotamase in Subjects With Cystic Fibrosis-Related Exocrine Pancreatic Insufficiency
Brief Title: SOLUTION: Study of Oral Liprotamase Unit-Matched Therapy Of Non-Porcine Origin in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN-EPI3331
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Exocrine Pancreatic Insufficiency; Cystic Fibrosis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis | interventions — liprotamase lipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liprotamase (Experimental): Individually-optimized dose to be administered orally
  Interventions: Drug: Liprotamase
- porcine (pig) PERT (Active Comparator): Individually-optimized dose to be administered orally
  Interventions: Drug: porcine (pig) PERT

INTERVENTIONS:
Drug: Liprotamase — oral, soluble, non-enterically coated, non-porcine, pancreatic enzyme replacement
  Arms: Liprotamase
Drug: porcine (pig) PERT — oral, enterically-coated, pancreatic replacement enzymes prepared from a porcine source
  Arms: porcine (pig) PERT

SUMMARY:
Liprotamase powder is a non-porcine, soluble and stable mixture of three digestive enzymes including lipase, protease, and amylase. The purpose of the present study is to provide additional efficacy and safety data compared to approved, porcine-derived, enterically-coated and encapsulated pancreatic enzyme replacement therapy. The primary efficacy endpoint of the study will be comparative efficacy measured as the change in the coefficient of fat absorption (CFA) in Cystic Fibrosis patients with exocrine pancreatic insufficiency (EPI).

Liprotamase is stable in stomach and digestive fluids allowing administration in a variety of convenient formulations and with a number of foods without enteric coating.

DETAILED DESCRIPTION:
Porcine derived enzymes are used for pancreatic enzyme replacement therapy in patients with cystic fibrosis (CF). Liprotamase is a biotechnology-derived enzyme replacement without enteric coating. This is an open-label, assessor blind, parallel group, multicenter, international trial to evaluate the noninferiority of liprotamase and pancrelipase in CF patients aged ≥7 years with pancreatic insufficiency. Subjects were randomized to liprotamase or pancrelipase, dose-matched to pre-study lipase doses. The lower bound of the 95% confidence interval (CI) for noninferiority was -15% for treatment difference in change from baseline coefficient of fat absorption (CFA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis based on presentation, genotype and/or sweat chloride
* Fecal elastase <100 mcg/g stool
* Minimum Coefficient of Fat (CFA) at screening while on stable PERT therapy
* Good nutritional status

Exclusion Criteria:

* History or diagnosis of fibrosing colonopathy
* Distal intestinal obstruction syndrome in 6 months prior to screening
* Receiving enteral tube feedings
* Chronic diarrheal illness unrelated to pancreatic insufficiency
* Liver abnormalities, or liver or lung transplant, or significant bowel resection
* Forced expiratory volume in 1 second (FEV1) <30%

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gangal, Study Director — Anthera Pharmaceuticals
Locations (54):
- United States (32):
  - Investigator Site 123, Long Beach, California
  - Investigator Site 107, Los Angeles, California
  - Investigator Site 114, Aurora, Colorado
  - Investigator Site 120, Gainesville, Florida
  - Investigator Site 102, Jacksonville, Florida
  - Investigator Site 130, Miami, Florida
  - Investigator Site 117, Orlando, Florida
  - Investigator Site 110, Atlanta, Georgia
  - Investigator Site 127, Chicago, Illinois
  - Investigator Site 109, Glenview, Illinois
  - Investigator Site 104, Indianapolis, Indiana
  - Investigator Site 105, Wichita, Kansas
  - Investigator Site 128, Lexington, Kentucky
  - Investigator Site 122, Louisville, Kentucky
  - Investigator Site 132, Portland, Maine
  - Investigator Site 124, Ann Arbor, Michigan
  - Investigator Site 126, East Lansing, Michigan
  - Investigator Site 134, Jackson, Mississippi
  - Investigator Site 135, Las Vegas, Nevada
  - Investigator Site 103, Cleveland, Ohio
  - Investigator Site 113, Toledo, Ohio
  - Investigator Site 101, Oklahoma City, Oklahoma
  - Investigator Site 136, Oklahoma City, Oklahoma
  - Investigator Site 119, Portland, Oregon
  - Investigator Site 106, Hershey, Pennsylvania
  - Investigator Site 115, Pittsburgh, Pennsylvania
  - Investigator Site 111, Dallas, Texas
  - Investigator Site 125, Fort Worth, Texas
  - Investigator Site 116, Houston, Texas
  - Investigator Site 121, Burlington, Vermont
  - Investigator Site 112, Richmond, Virginia
  - Investigator Site 129, Morgantown, West Virginia
- Investigator Site 133, Edmonton, Alberta, Canada
- Czechia (2):
  - Investigator Site 501, Brno
  - Investigator Site 502, Pilsen
- Hungary (5):
  - Investigator Site 305, Szeged, Csongrád megye
  - Investigator Site 303, Debrecen, Hajdú-Bihar
  - Investigator Site 302, Törökbálint, Pest County
  - Investigator Site 304, Mosdós, Somogy County
  - Investigator Site 301, Ajka, Veszprém megye
- Investigator Site 601, Jerusalem, Israel
- Poland (9):
  - Investigator Site 208, Bialystok
  - Investigator Site 203, Karpacz
  - Investigator Site 206, Lodz
  - Investigator Site 201, Lublin
  - Investigator Site 205, Lublin
  - Investigator Site 202, Rabka-Zdrój
  - Investigator Site 209, Rzeszów
  - Investigator Site 204, Sopot
  - Investigator Site 207, Warsaw
- Spain (4):
  - Investigator Site 403, Madrid
  - Investigator Site 401, Madrid
  - Investigator Site 402, Málaga
  - Investigator Site 404, Valencia

REFERENCES:
- [Derived] Somaraju URR, Solis-Moya A. Pancreatic enzyme replacement therapy for people with cystic fibrosis. Cochrane Database Syst Rev. 2020 Aug 5;8(8):CD008227. doi: 10.1002/14651858.CD008227.pub4. PMID 32761612

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liprotamase | Porcine (Pig) PERT
Started | 65 | 63
Completed | 47 | 59
Not Completed | 18 | 4
Not completed — Adverse Event | 3 | 0
Not completed — Lack of Efficacy | 4 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Undefined | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liprotamase | Porcine (Pig) PERT | Total
Number analyzed (Participants) | 65 | 63 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (8.54) | 21.0 (8.95) | 21.8 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 35 | 32 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 63 | 61 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Coefficient of fat absorption (CFA) [Mean (Full Range); unit: fat absorbed as percent of fat ingested] | 88.7 [80 to 98] | 89.4 [79 to 97] | 89.1 [79 to 98]
Coefficient of nitrogen absorption (CNA) [Mean (Full Range); unit: % of nitrogen ingested] | 96.9 [92 to 99] | 97.3 [94 to 99] | 97.1 [92 to 99]
pre-randomization enzyme dose [Mean (Full Range); unit: lipase units/kg/day] | 6299 [1190 to 9981] | 6264 [1692 to 9962] | 6282 [1190 to 9981]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Difference in Coefficient of Fat Absorption (CFA) Change From Baseline
Description: The primary endpoint evaluates the difference between treatment arms in change from baseline in coefficient of fat absorption (CFA). As such, descriptive statistics for individual treatment arms are not provided in this measure, but are reported in the secondary endpoints
Time Frame: Baseline, 7 weeks
Population: Analysis population evaluates all subjects who received at least one dose of study drug. Missing Visit 7 CFA values were multiply imputed using baseline CFA, baseline BMI, sex, age, acid suppression usage, and region.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change from baseline
Groups:
- Treatment Difference: analysed as LS mean difference in change in CFA from baseline for Liprotamase - Porcine enzymes
Arm/Group | Treatment Difference
Number analyzed (Participants) | 128
percent change from baseline | -11.852 [-16.0 to -7.7]

2. Secondary Outcome: Coefficient of Fat Absorption (CFA)
Description: Change from baseline in coefficient of fat absorption
Time Frame: Baseline, 7 weeks
Population: Analysis population evaluates observed case data without multiple imputation for missing values
Measure: Mean (Standard Deviation); unit: fat absorbed as % of fat ingested
Arm/Group | Liprotamase | Porcine (Pig) PERT
Number analyzed (Participants) | 53 | 62
fat absorbed as % of fat ingested | 76.5 (16.13) | 89.5 (5.84)

3. Secondary Outcome: Coefficient of Nitrogen Absorption (CNA)
Description: Change from baseline in coefficient of nitrogen absorption
Time Frame: Baseline, 7 weeks
Population: Analysis population evaluates observed case data without multiple imputation for missing values
Measure: Mean (Standard Deviation); unit: percent of nitrogen ingested
Arm/Group | Liprotamase | Porcine (Pig) PERT
Number analyzed (Participants) | 53 | 62
percent of nitrogen ingested | 95.8 (2.46) | 97.5 (1.21)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Liprotamase | Porcine (Pig) PERT
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/63
Serious Adverse Events (participants affected / at risk) | 7/65 | 6/63
Other Adverse Events (participants affected / at risk) | 41/65 | 38/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liprotamase (N=65) | Porcine (Pig) PERT (N=63)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liprotamase (N=65) | Porcine (Pig) PERT (N=63)
Infective pulmonary exacerbation (Infections and infestations) | 13 (13) | 17 (17)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other